CLINICAL TRIAL: NCT05827198
Title: Evaluating the Impact of Incremental Doses of a Sugar Replacer Blend on Gastrointestinal Tolerance in Candies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: INQUIS Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: KBE067 / INQ-2239
Record Dates: First submitted 2023-03-14; First posted 2023-04-24 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Gastrointestinal Tolerance; Healthy Population
Keywords: Sugar replacer; Gastrointestinal symptoms; BHD-BSS; GITQ; Acute

STUDY DESIGN:
Intervention Model Description: In a 4-way cross-over, there is a set of 4 balanced sequences to which participants will be randomly assigned (ABCD, BADC, CDAB, DCBA). Blocks of 2, 3, or 4 sets of sequences were randomly ordered to create a balanced sequence for n=60 participants. Orders will be assigned to participants in the order they attended for the first visit after being recruited.
Who Masked: Outcomes Assessor
Masking Description: The products will be labelled with a code and participants will not be informed which test meal is which. However, since the portion sizes of some of the treatments differ, some information about them may be available to participants and study coordinators; that is why we have termed the study "single blind". Single blinding will be achieved by identifying the treatments by code on the case report forms and in the database, so that those doing the statistical analysis and the study sponsor will be unaware of the treatment assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control sugar candies (Placebo Comparator): Control chewable candy made with sugar and provided at a dose of 50 g (corresponding to 2 servings)
  Interventions: Other: Low-sugar candies compared to regular sugar candies
- Test low sugar candies dose 1 (Active Comparator): low-sugar chewable candy containing Soluble Corn Fiber + Inulin + Erythritol provided at a dose of 50 g (corresponding to 2 servings)
  Interventions: Other: Low-sugar candies compared to regular sugar candies
- Test low sugar candies dose 2 (Active Comparator): 64% reduced sugar chewable candy containing Soluble Corn Fiber + Resistant wheat dextrins provided at a dose of 50 g (corresponding to 2 servings)
  Interventions: Other: Low-sugar candies compared to regular sugar candies
- Test low sugar candies dose 3 (Active Comparator): 82% reduced sugar chewable candy containing Soluble Corn Fiber + Resistant wheat dextrins provided at a dose of 50 g (corresponding to 2 servings)
  Interventions: Other: Low-sugar candies compared to regular sugar candies

INTERVENTIONS:
Other: Low-sugar candies compared to regular sugar candies — Acute intake

SUMMARY:
This study is a randomized, single-blind, crossover trial aiming at evaluating the gastrointestinal tolerance of a sugar replacer blend (inulin + soluble corn fiber + erythritol) at 3 different doses

DETAILED DESCRIPTION:
The study will have a randomized, single-blind, crossover design with 5 visits consisting of one screening visit and 4 study visits (3-14-day interval between the start of each visit) across 2-8 weeks. Participants will be randomized to a test sequence and will consume one control product and 3 test products made with the sugar replacer blend over the course of the study. At each visit, eligible participants will come to the lab between 8-11am, and ~1-2 hours after consuming their usual breakfast at home. After rating the severity of gastrointestinal symptoms, participants will consume one of the investigational products with a drink of water (250ml) and then be free to leave. The severity of 8 gastrointestinal symptoms (Abdominal bloating, Abdominal pain/discomfort, Gas/flatulence, Burping, Reflux (heartburn), Stomach rumbling (borborygmus), Nausea and Vomiting) will be rated at 2, 4, 6, 10 and 24 hours after starting to eat. Over the 24 hour period following consuming the investigational product a Bowel Habit Diary will be kept. For each bowel movement passed during the 24 hour period, participants will be asked to record: the time, if they had to strain, if they experienced discomfort, if they felt there was incomplete evacuation and the consistency of the stool rated using the using the Bristol Stool Scale (BSS).

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant, non-lactating, healthy individuals aged 18-55 years, inclusive
* BMI 18.5-32.0kg/m², inclusive
* No major illness, trauma or surgery requiring hospitalization within 3mo of the screening visit
* Ability to understand the study procedures and willing to provide informed consent to participate in the study
* Non-smokers or smokers who smoke <10 cigarettes/day and are willing not to change nicotine habits during the study period
* Willing to limit alcohol consumption to ≤3 standard drinks/d and ≤7 standard drinks/week during the study period
* Willing to refrain from any marijuana or hemp products during the study period
* Normal bowel habits (>2 bowel movements/week and <3 bowel movements per day)
* Consumes ≤4 servings/d of fruits and vegetables combined and ≤3 (women) or ≤4 (men) servings/d of whole grains using the definitions of "serving" .
* Participants must have a cell phone/tablet/computer and be willing and able to use it to collect study data
* Participants must be eligible to receive income in Canada and be covered by a health insurance plan such as OHIP
* Participants are willing to follow current COVID guidelines with respect to attending study visits

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria
* Chronic moderate to severe gastrointestinal symptoms
* Use of systemic antibiotics, antifungals or antiparasitics in the past 3 months and during the experimental period
* Use of medications, supplements, and products which may affect the results (laxative, anti-diarrhea, anti-constipation drugs, high fiber supplements)
* Individuals with any medical conditions or use of supplements or medications that increase risk to the subject or others or may affect the results, as judged by the Principal Investigator
* Unwillingness or inability to comply with the experimental procedures and to follow INQUIS safety guidelines
* Known intolerance, sensitivity, or allergy to any ingredients in the study test products
* Subject is currently participating or recently (within 30 days of screening) participated in a clinical trial involving long-term exposure (greater than 24 hours) to an investigational drug, nutritional supplement, or lifestyle modification

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-12 (Estimated); Primary Completion 2023-12-22 (Estimated); Study Completion 2024-01-27 (Estimated)

PRIMARY OUTCOMES:
Total Area Under the Curve (tAUC) of composite gastrointestinal Symptom score | tAUC between 0 and 24 hours
  total area under the curve (tAUC) of the composite GastroIntestinal symptom score (sum of the scores for the 8 GI symptoms). The score values can range from 0 up to 24 with the higher values showing the higher levels of symptoms (worse conditions).

SECONDARY OUTCOMES:
Total Area Under the Curve of each individual gastrointestinal symptom | tAUC between 0 and 24 hours
  Total Area Under the Curve of each of the individual 8 gastrointestinal symptoms. Each symptom range from 0 up to 3 with 3 showing the highest / worse condiiton of symptoms
Frequency of composite score > 1 at each time point | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Proportion of participants who have a composite GastoInestinal symptom score >1 (moderate-to-severe) at each time point. The composite score can range from 0 up to 24 with the higher values showing the higher levels of symptoms (worse conditions).
Frequency of Diarrhea within 24 hours | Evaluation performed over 24 hour after consumption of study products
  Proportion of participants with diarrhea, defined as 3 or more type 6 or 7 stools (based on the BSS) within the 24 hour period after consumption of the study products
Maximum score and time for maximum score for each gastrointestinal symptom | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  For each individual GI symptom: the proportion of participants reporting any (score>0) or moderate/severe (score >1) at each time point, the maximum detected score (which can range from 0 up to 3) and the time of the maximum score
Number of bowel movements | Evaluation performed over 24 hour after consumption of study products
  Number of bowel movements over the 24 hours
straining during bowel movement | Evaluation performed over 24 hour after consumption of study products
  Proportion of participants having to strain or not
discomfort during bowel movement | Evaluation performed over 24 hour after consumption of study products
  Proportion of participants having discomfort or not
incomplete evacuation | Evaluation performed over 24 hour after consumption of study products
  Proportion of participants declaring incomplete evacuation or not
Stool consistency based on britol stool scale | Evaluation performed over 24 hour after consumption of study products
  mean stool consistency on Bristol Stool Scale (BSS). The scale provide values from 1 to 7 depending on the type of stool with 1 being the driest stools and 7 the most liquid one.

CONTACTS AND LOCATIONS:
Locations (1):
- Inquis Clinical Research, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No